CLINICAL TRIAL: NCT03412110
Title: Assessment & Feasibility of an Electronic Post-Symptoms Evaluation
Brief Title: (MIST2)-Part2: AEs Following DC Care at DC Teaching Clinic: Electronic
Acronym: MIST2
Status: Completed | Type: Observational
Sponsor: Parker University (Other)
Collaborators: Canadian Memorial Chiropractic College (Other); University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Parker17_002
Record Dates: First submitted 2018-01-17; First posted 2018-01-26 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Patient Safety; Manipulation, Spinal
Keywords: chiropractic; SMT; Active surveillance reporting system

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: active surveillance: electronic platform — Provides a structure to systematically gather adverse event information from healthcare providers and sometimes directly from patients.

SUMMARY:
This study aims to compare different ways to establish severity from patients reporting a new or worsening symptom (adverse event) following a chiropractic treatment at a teaching clinic using an electronic platform.

DETAILED DESCRIPTION:
Healthcare systems acknowledge the importance of patient safety including the reduction of preventable adverse events (AE). For healthcare providers who perform spinal manipulation therapy (SMT), the investigation of AEs remains in its infancy for several reasons including finding a reporting system that accurately collects AEs information, varied descriptions of AE's severity and occurrence frequency and the variable natural history of musculoskeletal conditions treated by SMT. Together, these factors act together to conspire against the implementation of systematic changes in SMT application that would result in improved patient care and safety.

In addition, it is vital that patient safety training initiates at the start of a healthcare worker's career. This pilot active surveillance study was designed to assess the feasibility of collecting data with an electronic platform for patients' self-report of symptom changes as well as interns' report at a chiropractic teaching clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the Parker University Wellness Clinic
* Agreed to participate

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Each supervising faculty clinician in the Parker Wellness Clinic had data collected from interested patients during a pre-specified one week period of time.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
patient - report of an adverse event | Up to 7 days post treatment - Day 0-7
  as any unfavorable sign, symptom or disease temporarily associated with the treatment, whether or not caused by the treatment, specifically any worsened or new symptom reported by the patient up to one week after care
intern - report of an adverse event | Immediate after treatment - Day 0
  as any unfavorable sign, symptom or disease temporarily associated with the treatment, whether or not caused by the treatment, specifically any worsened or new symptom reported by the intern immediately following care

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Pohlman, DC, MS, Principal Investigator — Parker University
Locations (1):
- Parker University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Informed Consent Form: Patient Consent Form (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03412110/ICF_000.pdf
  • Informed Consent Form: Clinician/ Student Consent Form (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03412110/ICF_001.pdf